CLINICAL TRIAL: NCT04672096
Title: Basic Assessment of Safety and Minimally Invasive Stimulation Via Injectrode
Acronym: BASMATI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuronoff, Inc (Industry)
Collaborators: Ohio Pain Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NCP-01
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-11

CONDITIONS: Chronic Lower Limb Pain
Keywords: Electrode; Injectable Electrode; Injectrode; Medical Device Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Neuronoff BASMATI Injectrode (Experimental): Subjects will be provided with the placement of an Injectrode insert. The maximal placement duration will be 28 days.
  Interventions: Device: Neuronoff BASMATI Injectrode

INTERVENTIONS:
Device: Neuronoff BASMATI Injectrode — The 28 day temporary placement of a Basmati Injectrode does not result in unexpected levels of inflammation or encapsulation.
  Other Names: Injectrode; BASMATI Injectrode

SUMMARY:
The objectives of this non-significant risk (NSR) study are to evaluate the safety of the short term placement of the Basmati Injectrode for up to 28 days and the efficacy of conducting electrical current to stimulate subcutaneous nerves on the explant date just prior to explant.

DETAILED DESCRIPTION:
This was a prospective, single-center, single-arm, non-randomized study design. A sample of 10 study participants were enrolled into the study, and provided with the placement of a Basmati Injectrode insert with a maximal placement duration of up to 28 days. Subjects who were selected to participate in the trial were healthy volunteers adults with ages 18 years and older without any preexisting condition indicated for treatment. Each subject was followed during the trial period of approximately 45+/-2 days.

ELIGIBILITY:
Inclusion Criteria:

* Sign a valid, Institutional Review Board (IRB)-approved informed consent form (ICF) and understand the study requirements.
* Be 18 years of age or older when written informed consent is obtained.
* Be in good physical and mental health as assessed by a general practitioner.
* Be able to tolerate electrical stimulation (TENS).
* Be willing and able to understand and comply with all study-related procedures during the course of the study.

Exclusion Criteria:

* Have a cognitive impairment or exhibit any characteristic that would limit the study candidate's ability to completely understand and sign a valid, IRB-approved informed consent form.
* Have a positive pregnancy test (conducted during enrollment).
* Have a positive Allergic reactivity to Gold skin test (conducted during enrollment).
* Show symptoms indicative for Covid19 as assessed during enrollment.
* Have a skin condition at the planned surgical location.
* Have a blood coagulation disorder or other indication with the potential to impact the study biocompatibility data in unpredictable ways.
* Have a medical condition that is a contraindication for minimally invasive surgery.
* Be implanted with a cardiac defibrillator or pump.
* Have a history of cardiac arrhythmia with hemodynamic instability
* Be implanted with a neurostimulator.
* Have any active electrical implant of any other kind.
* Have metal implants (particularly in hip).
* Have active infection.
* Have allodynia.
* Take regular use of antiplatelet medications (e.g. aspirin, ticlopidine (Ticlid), clopidogrel (Plavix), tirofiban (Aggrastat) or eptifibatide (Integrilin)).
* Have untreated drug habituation or dependence.
* Have uncontrolled seizures (averaging > 2 seizures per month).
* Currently require, or be likely to require, diathermy and/or MRI during study duration.
* Have a history of adverse reactions to local anesthetics (e.g. lidocaine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amol Soin, MD, Principal Investigator — Ohio Pain Clinic
Locations (1):
- Ohio Pain Clinic, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Neuronoff BASMATI Injectrode: This group was evaluated to 1) assess tissue responses and, on the last day just prior to explant, 2) collect data describing the quality of the electrical interfacing with the Injectrode from outside of the body, as well as with subcutaneous sensory nerves surrounding the Injectrode insert.
Period: Overall Study
Arm/Group | Neuronoff BASMATI Injectrode
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Neuronoff BASMATI Injectrode: See Inclusion/Exclusion Criteria
Arm/Group | Neuronoff BASMATI Injectrode
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety - Number of Participants With Device-Related Adverse Events & Histological Analysis
Description: Primary measures of device safety included verification of the absence of unexpected inflammation and minimization of excessive encapsulation around the Injectrode as verified by cell staining and pathohistological analysis.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Neuronoff BASMATI Injectrode: Subjects will be provided with the placement of an Injectrode insert. The maximal placement duration will be 28 days. On the day of explant, stimulation of the Injectrode will occur for approximately 30 minutes.
  Neuronoff BASMATI Injectrode: The 28 day temporary placement of a Basmati Injectrode does not result in unexpected levels of inflammation or encapsulation.
Arm/Group | Neuronoff BASMATI Injectrode
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Neuronoff BASMATI Injectrode
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuronoff BASMATI Injectrode (N=10)
Shingles - Unrelated (Skin and subcutaneous tissue disorders) | 1 (1) — Subject presented with shingles, unrelated to subject device or procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT04672096/Prot_000.pdf
  • Informed Consent Form (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT04672096/ICF_001.pdf